CLINICAL TRIAL: NCT02138916
Title: Randomised, Double-blind, 56 Week Placebo-controlled, Parallel Group, Multicentre, Phase 3 Study to Evaluate the Efficacy and Safety of 2 Doses of Benralizumab in Patients With Moderate to Very Severe COPD With a History of Exacerbations
Brief Title: Benralizumab Efficacy in Moderate to Very Severe Chronic Obstructive Pulmonary Disease (COPD) With Exacerbation History
Acronym: GALATHEA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3251C00003
Record Dates: First submitted 2014-03-26; First posted 2014-05-15 (Estimated); Results first posted 2019-06-13 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Moderate to Very Severe Chronic Obstructive Pulmonary Disease
Keywords: Obstructive Lung Diseases; Chronic Obstructive Pulmonary Disease; Lung Disease; Bronchial Diseases; COPD Exacerbation; Respiratory Tract Diseases
MeSH Terms: conditions — Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive; Lung Diseases; Bronchial Diseases; Respiratory Tract Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Benralizumab Arm A (Experimental): Benralizumab administered subcutaneously
  Interventions: Drug: Benralizumab Arm A
- Benralizumab Arm B (Experimental): Benralizumab administered subcutaneously
  Interventions: Drug: Benralizumab Arm B
- Placebo (Placebo Comparator): Placebo administered subcutaneously
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Benralizumab Arm A — Benralizumab subcutaneously on study week 0 until study week 48 inclusive
  Arms: Benralizumab Arm A
Drug: Benralizumab Arm B — Benralizumab subcutaneously on study week 0 until study week 48 inclusive
  Arms: Benralizumab Arm B
Drug: Placebo — Placebo subcutaneously on study week 0 until study week 48 inclusive
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine if benralizumab reduces COPD exacerbation rate in symptomatic patients with moderate to very severe COPD who are receiving standard of care therapies

ELIGIBILITY:
Inclusion Criteria:1.Informed consent. 2.Subjects 40-85 y.o. 3.Moderate to very severe COPD with Post Bronchodilator (BD) FEV1>20% and ≤65%. 4.≥2 moderate or ≥1 severe COPD exacerbation(s) required treatment or hospitalization within 2-52 weeks prior to Visit1. 5. Modified Medical Research Council (mMRC) score ≥1 at Visit 1. 6.Treatment with double or triple therapy throughout the year prior to Visit 1, constant 2 weeks prior to Visit 1. 7.Tobacco history of ≥10 pack-years. 8.Women of childbearing potential must use a highly effective form of birth control from Visit 1 until 16 weeks after their last dose, and negative serum pregnancy test result at Visit 1. 9.Male subjects who are sexually active must be surgically sterile one year prior to Visit 1 or use an adequate method of contraception from the first Investigational Product (IP) dose until 16 weeks after their last dose. 10.Compliance with maintenance therapy during run-in ≥70%. 11. Blood eosinophils due to subject's stratification and cap for blood eosinophil levels.When any eosinophil cohort is full, subjects in the completed cohort will not be randomised and will be withdrawn from the study. Exclusion criteria: 1. Clinically important pulmonary disease other than COPD or another diagnosed pulmonary or systemic disease associated with elevated peripheral eosinophil counts.

2. Any disorder or major physical impairment that is not stable by Investigator opinion and/or could affect: - subject safety-study findings or their interpretation or subject's ability to complete the entire study duration.

3. Unstable ischemic heart disease, arrhythmia, cardiomyopathy, or other relevant cardiovascular disorder that in Investigator's judgment may put the patient at risk or negatively affect the study outcome.

4. Treatment with systemic corticosteroids and/or antibiotics, and/or hospitalization for a COPD exacerbation within 2 weeks prior to Visit1 or during the enrolment and run-in period.

5. Acute upper or lower respiratory infection requiring antibiotics or antiviral medication within 2 weeks prior to Visit1or during the enrolment and run-in period.

6. Pneumonia within 8 weeks prior to Visit1 or during the enrolment and run-in period.

7. Pregnant, breastfeeding, or lactating women. 8. Risk factors for pneumonia 9. History of anaphylaxis to any other biologic therapy. 10. Long term oxygen therapy with signs and/or symptoms of cor pulmonale, right ventricular failure.

11. Use of immunosuppressive medication within 2 weeks prior to Visit1 and/or during the enrolment and run-in period.

12. Receipt of any investigational non-biologic product within 30 days or 5 half-lives prior to Visit 1.

13. Evidence of active tuberculosis (TB) without an appropriate course of treatment.

14. Lung volume reduction surgery within the 6 months prior to Visit 1. History of partial or total lung resection (single lobe or segmentectomy is acceptable).

15. Asthma as a primary or main diagnosis according to the Global Initiative for Asthma (GINA) guidelines or other accepted guidelines.

16. Previous treatment with benralizumab. 17. Helminth parasitic infection diagnosed within 24 weeks prior to Visit 1.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1656 (Actual)
Dates: Start 2014-06-13 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Criner, MD, Principal Investigator — Temple University School of Medicine, 3401 North Broad Street, Suite 745 PP, Philadelphia, PA 19140
Locations (338):
- United States (117):
  - Research Site, Andalusia, Alabama
  - Research Site, Birmingham, Alabama
  - Research Site, Dothan, Alabama
  - Research Site, Jasper, Alabama
  - Research Site, Little Rock, Arkansas
  - Research Site, Beverly Hills, California
  - Research Site, Gold River, California
  - Research Site, Huntington Beach, California
  - Research Site, Huntington Park, California
  - Research Site, Lakewood, California
  - Research Site, Lomita, California
  - Research Site, Newport Beach, California
  - Research Site, Palm Desert, California
  - Research Site, Palo Alto, California
  - Research Site, Riverside, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Santa Ana, California
  - Research Site, Thousand Oaks, California
  - Research Site, Torrance, California
  - Research Site, New Haven, Connecticut
  - Research Site, Waterbury, Connecticut
  - Research Site, Boynton Beach, Florida
  - Research Site, Brandon, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Loxahatchee Groves, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Springs, Florida
  - Research Site, Orlando, Florida
  - Research Site, Panama City, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Sebring, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Vero Beach, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Calhoun, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Duluth, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Eagle, Idaho
  - Research Site, Aurora, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, Michigan City, Indiana
  - Research Site, Valparaiso, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, Fort Mitchell, Kentucky
  - Research Site, Hazard, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Columbia, Maryland
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Farmington Hills, Michigan
  - Research Site, Rochester, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Saint Charles, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Summit, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Bronxville, New York
  - Research Site, Brooklyn, New York
  - Research Site, Buffalo, New York
  - Research Site, Fayetteville, New York
  - Research Site, New York, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Elizabeth City, North Carolina
  - Research Site, Gastonia, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Mount Airy, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Bend, Oregon
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Altoona, Pennsylvania
  - Research Site, Erie, Pennsylvania
  - Research Site, Jefferson Hills, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Wyomissing, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Columbia, South Carolina
  - Research Site, Gaffney, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Old Point Station, South Carolina
  - Research Site, Rock Hill, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Chattanooga, Tennessee
  - Research Site, Franklin, Tennessee
  - Research Site, Hendersonville, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Austin, Texas
  - Research Site, Boerne, Texas
  - Research Site, Frisco, Texas
  - Research Site, Galveston, Texas
  - Research Site, Houston, Texas
  - Research Site, McAllen, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Tyler, Texas
  - Research Site, Midvale, Utah
  - Research Site, Provo, Utah
  - Research Site, Richmond, Virginia
  - Research Site, Richland, Washington
- Austria (7):
  - Research Site, Feldkirch
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Vienna
  - Research Site, Wels
- Canada (13):
  - Research Site, Calgary, Alberta
  - Research Site, Sherwood Park, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Ajax, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Grimsby, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Pointe-Claire, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Trois-Rivières, Quebec
  - Research Site, Saskatoon, Saskatchewan
- Czechia (9):
  - Research Site, Jindřichův Hradec
  - Research Site, Karlovy Vary
  - Research Site, Kralupy nad Vltavou
  - Research Site, Mladá Boleslav
  - Research Site, Olomouc
  - Research Site, Prague
  - Research Site, Rokycany
  - Research Site, Strakonice
  - Research Site, Teplice
- Germany (13):
  - Research Site, Bamberg
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Frankfurt
  - Research Site, Frankfurt am Main
  - Research Site, Geesthacht
  - Research Site, Hamburg
  - Research Site, Leipzig
  - Research Site, Marburg
  - Research Site, Neu-Isenburg
  - Research Site, Rodgau-Dudenhofen
  - Research Site, Teuchern
  - Research Site, Witten
- Hungary (13):
  - Research Site, Balassagyarmat
  - Research Site, Budapest
  - Research Site, Edelény
  - Research Site, Farkasgyepü
  - Research Site, Gödöllő
  - Research Site, Hajdúnánás
  - Research Site, Hatvan
  - Research Site, Mátraháza
  - Research Site, Miskolc
  - Research Site, Pécs
  - Research Site, Százhalombatta
  - Research Site, Szeged
  - Research Site, Székesfehérvár
- Italy (10):
  - Research Site, Bolzano
  - Research Site, Catania
  - Research Site, Ferrara
  - Research Site, Genova
  - Research Site, Orbassano
  - Research Site, Palermo
  - Research Site, Parma
  - Research Site, Pavia
  - Research Site, Pisa
  - Research Site, Tradate
- Japan (60):
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Fukuyama-shi
  - Research Site, Higashiibaraki-gun
  - Research Site, Himeji-shi
  - Research Site, Hirosaki-shi
  - Research Site, Iwata-shi
  - Research Site, Izumo-shi
  - Research Site, Joyo-shi
  - Research Site, Kagoshima
  - Research Site, Kasuga-shi
  - Research Site, Kasugai-shi
  - Research Site, Kawaguchi-shi
  - Research Site, Kawasaki-shi
  - Research Site, Kiryu-shi
  - Research Site, Kishiwada-shi
  - Research Site, Kitakami-shi
  - Research Site, Kobe
  - Research Site, Kochi
  - Research Site, Kodaira-shi
  - Research Site, Kokubunji-shi
  - Research Site, Koshi-shi
  - Research Site, Kuki-shi
  - Research Site, Kumamoto
  - Research Site, Kurashiki-shi
  - Research Site, Kurume-shi
  - Research Site, Kyoto
  - Research Site, Matsue
  - Research Site, Matsumoto-shi
  - Research Site, Matsusaka-shi
  - Research Site, Meguro-ku
  - Research Site, Mizunami-shi
  - Research Site, Morioka
  - Research Site, Nagaoka-shi
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Obihiro-shi
  - Research Site, Ohota-ku
  - Research Site, Ota-shi
  - Research Site, Saiki-shi
  - Research Site, Sakaide-shi
  - Research Site, Sakaishi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Seto-shi
  - Research Site, Shinagawa-ku
  - Research Site, Shinjuku-ku
  - Research Site, Takamatsu
  - Research Site, Takatsuki-shi
  - Research Site, Toon-shi
  - Research Site, Toshima-ku
  - Research Site, Ube-shi
  - Research Site, Ueda-shi
  - Research Site, Uji-shi
  - Research Site, Urasoe-shi
  - Research Site, Uruma
  - Research Site, Yachiyo-shi
  - Research Site, Yakushi
  - Research Site, Yanagawa-shi
  - Research Site, Yokohama
- Netherlands (6):
  - Research Site, Breda
  - Research Site, Eindhoven
  - Research Site, Heerlen
  - Research Site, Horn
  - Research Site, Nijmegen
  - Research Site, Zwolle
- Poland (19):
  - Research Site, Bydgoszcz
  - Research Site, Dobre Miasto
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Kościan
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Mrągowo
  - Research Site, Mrozy
  - Research Site, Olsztyn
  - Research Site, Proszowice
  - Research Site, Radom
  - Research Site, Ruda Śląska
  - Research Site, Rzeszów
  - Research Site, Tarnów
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Zakopane
- Romania (7):
  - Research Site, Bragadiru
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Constanța
  - Research Site, Deva
  - Research Site, Iași
  - Research Site, Timișoara
- Russia (23):
  - Research Site, Chelyabinsk
  - Research Site, Ivanovo
  - Research Site, Izhevsk
  - Research Site, Kazan'
  - Research Site, Kemerovo
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Penza
  - Research Site, Perm
  - Research Site, Pskov
  - Research Site, Pyatigorsk
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Smolensk
  - Research Site, Tomsk
  - Research Site, Ufa
  - Research Site, Ulyanovsk
  - Research Site, Vladikavkaz
  - Research Site, Vladimir
  - Research Site, Volgograd
  - Research Site, Yekaterinburg
- South Africa (6):
  - Research Site, Bloemfontein
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, eManzimtoti
  - Research Site, Gauteng
  - Research Site, Middelburg
- South Korea (4):
  - Research Site, Bucheon-si
  - Research Site, Daegu
  - Research Site, Seoul
  - Research Site, Wŏnju
- Spain (9):
  - Research Site, Alicante
  - Research Site, Badalona(Barcelona)
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Palma de Mallorca
  - Research Site, Sabadell (Barcelona)
  - Research Site, Santander
  - Research Site, Valencia
- Switzerland (5):
  - Research Site, Basel
  - Research Site, Biel
  - Research Site, Gossau
  - Research Site, Liestal
  - Research Site, Sankt Gallen
- United Kingdom (17):
  - Research Site, Aberdeen
  - Research Site, Birmingham
  - Research Site, Bradford
  - Research Site, Cambridge
  - Research Site, Chertsey
  - Research Site, Edinburgh
  - Research Site, Glasgow
  - Research Site, LE3 9QP
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Newcastle-under-Lyme
  - Research Site, Oxford
  - Research Site, Plymouth
  - Research Site, Southampton
  - Research Site, Wishaw
  - Research Site, Wolverhampton

REFERENCES:
- [Derived] Criner GJ, Celli BR, Singh D, Agusti A, Papi A, Jison M, Makulova N, Shih VH, Brooks L, Barker P, Martin UJ, Newbold P. Predicting response to benralizumab in chronic obstructive pulmonary disease: analyses of GALATHEA and TERRANOVA studies. Lancet Respir Med. 2020 Feb;8(2):158-170. doi: 10.1016/S2213-2600(19)30338-8. Epub 2019 Sep 28. PMID 31575508
- [Derived] Criner GJ, Celli BR, Brightling CE, Agusti A, Papi A, Singh D, Sin DD, Vogelmeier CF, Sciurba FC, Bafadhel M, Backer V, Kato M, Ramirez-Venegas A, Wei YF, Bjermer L, Shih VH, Jison M, O'Quinn S, Makulova N, Newbold P, Goldman M, Martin UJ; GALATHEA Study Investigators; TERRANOVA Study Investigators. Benralizumab for the Prevention of COPD Exacerbations. N Engl J Med. 2019 Sep 12;381(11):1023-1034. doi: 10.1056/NEJMoa1905248. Epub 2019 May 20. PMID 31112385
- See also: Clinical Study protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2562&filename=Galathea_CSP_and_last_amendment_Redacted.pdf
- See also: Statistical Analysis Plan (SAP) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2562&filename=D3251C00003_Statistical_Analysis_Plan_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1656 patients randomized to Benralizumab 30 mg, Benralizumab 100 mg, or Placebo. All randomized patients were treated. 554 (33.5%) were randomized to Benralizumab 30 mg, 552 (33.3%) were randomized to Benralizumab 100 mg, and 550 (33.2%) were randomized to Placebo.
Groups:
- Benralizumab 30 mg; Benralizumab 100 mg; Placebo: Every 8 weeks administered subcutaneously
Period: Overall Study
Arm/Group | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Started | 554 | 552 | 550
Completed | 497 | 492 | 491
Not Completed | 57 | 60 | 59
Not completed — eg., meds change, lack of efficacy, etc. | 6 | 9 | 7
Not completed — Death | 14 | 11 | 12
Not completed — Withdrawal by Subject | 27 | 31 | 32
Not completed — Study specific withdrawal criteria | 0 | 0 | 1
Not completed — incorrect enrolment | 1 | 1 | 0
Not completed — Severe non-compliance | 1 | 2 | 1
Not completed — Lost to Follow-up | 4 | 2 | 3
Not completed — Adverse Event | 4 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Benralizumab 30 mg | Benralizumab 100 mg | Placebo | Total
Number analyzed (Participants) | 554 | 552 | 550 | 1656
Age, Continuous [Mean (Standard Deviation); unit: Year] — Population: Full analysis set
  Year | 65.9 (7.77) | 65.3 (8.05) | 65.2 (8.22) | 65.5 (8.01)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Full analysis set
  Participants
    Female | 172 | 180 | 175 | 527
    Male | 382 | 372 | 375 | 1129
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Full analysis set
  Participants
    White | 496 | 493 | 488 | 1477
    Black or African American | 4 | 11 | 10 | 25
    Asian | 48 | 46 | 46 | 140
    Other | 6 | 2 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Annual COPD Exacerbation Rate Over 56 Weeks Treatment Comparison for Patients With Baseline EOS>=220/uL
Description: A COPD exacerbation is defined by symptomatic worsening of COPD requiring:
  * Use of systemic corticosteroids for at least 3 days; a single depot injectable dose of corticosteroids will be considered equivalent to a 3-day course of systemic corticosteroids; and/or
  * Use of antibiotics; and/or
  * An inpatient hospitalization or death due to COPD Annual COPD exacerbation rate is the number of exacerbations per year. Its raw rate is calculated by number of exacerbations divided by the treatment period and then normalized to an annual rate, and is estimated by negative binomial model. Rate ratio between two treatment groups is also estimated through this model.
Time Frame: From first IP to week 56
Population: Full analysis set with baseline EOS>=220/uL
Measure: Least Squares Mean (95% Confidence Interval); unit: Exacerbations per year
Arm/Group | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 382 | 379 | 359
Exacerbations per year | 1.19 [1.04 to 1.36] | 1.03 [0.9 to 1.19] | 1.24 [1.08 to 1.42]
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.6490, Negative binomial; Model includes treatment group, EOS cohort, region, background therapy, number of exacerbations in the previous year; Rate ratio = 0.96, 95% CI 2-sided [0.8 to 1.15]
Statistical Analysis 2: Comparison: Benralizumab 100 mg vs Placebo; Test type: Superiority; p = 0.0525, Negative binomial; Model includes treatment group, EOS cohort, region, background therapy, number of exacerbations in the previous year; Risk Ratio (RR) = 0.83, 95% CI 2-sided [0.69 to 1.00]

2. Secondary Outcome: Annual COPD Exacerbation Rate Over 56 Weeks Treatment Comparison for Patients With Baseline EOS<220/uL
Description: as for outcome 1
Time Frame: From first IP to week 56
Population: Full analysis set with baseline EOS<220/uL
Measure: Least Squares Mean (95% Confidence Interval); unit: Exacerbations per year
Arm/Group | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 172 | 173 | 191
Exacerbations per year | 1.4 [1.19 to 1.64] | 1.32 [1.12 to 1.56] | 1.30 [1.11 to 1.52]
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.5236, Negative binomial; Model includes treatment group, region, number of exacerbations in the previous year; Risk Ratio (RR) = 1.07, 95% CI 2-sided [0.86 to 1.34]
Statistical Analysis 2: Comparison: Benralizumab 100 mg vs Placebo; Test type: Superiority; p = 0.8812, Negative binomial; Model includes treatment group, EOS cohort, region, number of exacerbations in the previous year; Risk Ratio (RR) = 1.02, 95% CI 2-sided [0.82 to 1.27]

3. Secondary Outcome: Mean Change From Baseline to Week 56 in Pre-bronchodilator FEV1 (L) Value for Patients With Baseline EOS>=220/uL
Description: Pre-bronchodilator FEV1 (L) is collected at Weeks 0, 4, 8, 16, 24, 32, 40, 48, and 56. Baseline is the last non-missing value with quality (acceptable or borderline quality grade) prior to the first dose of study treatment.
Time Frame: First IP up to end of treatment Week 56
Population: Full analysis set, baseline EOS>=220/uL
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 329 | 326 | 317
Liter | 0.014 (0.282) | 0.031 (0.294) | 0.010 (0.275)
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.7550, Mixed Models Analysis; Model includes treatment group, baseline FEV1 value, EOS cohort, region, background therapy, visit, and treatment by visit interaction; Mean Difference (Final Values) = 0.007, 95% CI 2-sided [-0.035 to 0.048]
Statistical Analysis 2: Comparison: Benralizumab 100 mg vs Placebo; Test type: Superiority; p = 0.3285, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.021, 95% CI 2-sided [-0.021 to 0.062]

4. Secondary Outcome: Mean Change From Baseline in SGRQ Total Score for Patients With Baseline EOS>=220/uL
Description: SGRQ is from 50-item PRO instrument. The SGRQ total score is expressed as a percentage of overall impairment, in which 100% means the worst possible health status and 0 indicates the best possible health status.
Time Frame: First IP up to Week 56
Population: Full analysis set, baseline EOS>=220/uL
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 338 | 331 | 317
Percentage | -5.025 (14.677) | -6.723 (15.723) | -3.913 (15.039)
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.2906, Mixed Models Analysis; Model includes treatment group, baseline SGRQ score, EOS cohort, region, background therapy, visit, and treatment by visit interaction; Mean Difference (Final Values) = -1.011, 95% CI 2-sided [-2.887 to 0.865]
Statistical Analysis 2: Comparison: Benralizumab 100 mg vs Placebo; Test type: Superiority; p = 0.0264, Mixed Models Analysis; [statistical method as in outcome 4, analysis 1]; Mean Difference (Final Values) = -2.136, 95% CI 2-sided [-4.020 to -0.251]

5. Secondary Outcome: Mean Change From Baseline in CAT Total Score for Patients With Baseline EOS>=220/uL
Description: CAT is an 8-item PRO developed to measure the impact of COPD on health status. The instrument uses semantic differential six-point response scales. A CAT total score is the sum of item responses. Score ranges from 0 to 40 with higher scores indicative of greater COPD impact on health status.
Time Frame: First IP up to Week 56
Population: Full analysis set, baseline EOS>=220/uL
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 338 | 335 | 319
Score on a scale | -1.50 (6.89) | -2.43 (6.34) | -1.22 (6.53)
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.6782, Mixed Models Analysis; Model includes treatment group, baseline CAT total score, EOS cohort, region, background therapy, visit, and treatment by visit interaction; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-1.08 to 0.70]
Statistical Analysis 2: Comparison: Benralizumab 100 mg vs Placebo; Test type: Superiority; p = 0.0753, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.81, 95% CI 2-sided [-1.70 to 0.08]

6. Secondary Outcome: Mean Change From Baseline in E-RS: COPD Total Score for Patients With Baseline EOS>=220/uL
Description: The E-RS: COPD is an 11-item PRO developed to evaluate the severity of respiratory symptoms of COPD. Summation of E-RS: COPD item responses produces a total score ranging from 0 to 40, with higher scores indicating greater severity.
Time Frame: First IP up to Week 56
Population: Full analysis set, baseline EOS>=220/uL
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 324 | 328 | 295
Score on a scale | -1.085 (5.273) | -1.354 (5.599) | -0.504 (5.674)
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.0889, Mixed Models Analysis; Model includes treatment group, baseline total score, EOS cohort, region, background therapy, visit, and treatment by visit interaction; Mean Difference (Final Values) = -0.585, 95% CI 2-sided [-1.260 to 0.089]
Statistical Analysis 2: Comparison: Benralizumab 100 mg vs Placebo; Test type: Superiority; p = 0.0413, Mixed Models Analysis; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.703, 95% CI 2-sided [-1.378 to -0.028]

7. Secondary Outcome: Mean Change From Baseline in Total Rescue Medication Use (Number of Puffs Per Day) for Patients With Baseline EOS>=220/uL
Description: The number of rescue medication inhalations and nebulizer treatments taken are recorded by the patient in the eDiary twice daily. Total rescue medication use is the sum of daytime and night-time use.
Time Frame: First IP up to Week 56
Population: Full analysis set, baseline EOS>=220/uL
Measure: Mean (Standard Deviation); unit: Puffs/day
Arm/Group | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 321 | 322 | 291
Puffs/day | -0.05 (3.21) | -0.27 (2.71) | 0.29 (3.03)
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.0728, Mixed Models Analysis; Model includes treatment group, baseline rescue med. use, EOS cohort, region, background therapy, visit, and treatment by visit interaction; Mean Difference (Final Values) = -0.348, 95% CI 2-sided [-0.728 to 0.032]
Statistical Analysis 2: Comparison: Benralizumab 100 mg vs Placebo; Test type: Superiority; p = 0.0121, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -0.487, 95% CI 2-sided [-0.868 to -0.107]

8. Secondary Outcome: Mean Change From Baseline in Proportion of Nights Awakenings Due to Respiratory Symptoms for Patients With Baseline EOS>=220/uL
Description: Change from baseline to week 56 in proportion of nights awakenings due to respiratory symptoms.
Time Frame: First IP up to Week 56
Population: Full analysis set, baseline EOS>=220/uL
Measure: Mean (Standard Deviation); unit: Proportion of nights
Arm/Group | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 325 | 323 | 297
Proportion of nights | -0.088 (0.310) | -0085 (0.283) | -0.049 (0.307)
Statistical Analysis 1: Comparison: Benralizumab 30 mg; Test type: Superiority; p = 0.0235, Mixed Models Analysis; Model includes treatment group, baseline prop. of nights awakens., EOS cohort, region, background therapy, visit, and treatment by visit interaction; Mean Difference (Final Values) = -0.041, 95% CI 2-sided [-0.077 to -0.006]
Statistical Analysis 2: Comparison: Benralizumab 100 mg; Test type: Superiority; p = 0.0158, Mixed Models Analysis; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -0.044, 95% CI 2-sided [-0.080 to -0.008]

9. Secondary Outcome: Number of Participants by Number of COPD Exacerbations Based on EXACT-PRO for Patients With Baseline EOS>=220/uL
Description: The EXACT-PRO is a 14-item PRO instrument developed to assess the frequency, severity and duration of COPD exacerbations. Respondents are instructed to complete the electronic diary (eDiary) each evening just prior to bedtime and to answer the questions while onsidering their experiences "today". The daily EXACT-PRO total score has a range of 0-100 with higher scores indicative of greater severity. Exacerbation event frequency is calculated by comparing the baseline with daily total scores. An increase in EXACT-PRO total score ≥9 for 3 days or ≥12 for 2 days indicate an exacerbation event has occurred.
Time Frame: Immediately following first IP up to week 56
Population: Full analysis set, EOS>=220/uL
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 382 | 378 | 358
Participants
  0 | 180 | 184 | 179
  1 | 101 | 103 | 99
  2 | 42 | 49 | 34
  3 | 25 | 14 | 15
  4 | 17 | 13 | 14
  5 | 5 | 6 | 5
  6 | 4 | 4 | 2
  7 | 6 | 1 | 5
  8 | 1 | 1 | 4
  9 | 1 | 2 | 1
  10 | 0 | 1 | 0

10. Secondary Outcome: Severity of EXACT-PRO for Patients With Baseline EOS>=220/uL
Description: The EXACT-PRO is a 14-item PRO instrument developed to assess the frequency, severity and duration of COPD exacerbations. Respondents are instructed to complete the electronic diary (eDiary) each evening just prior to bedtime and to answer the questions while onsidering their experiences "today". The daily EXACT-PRO total score has a range of 0-100 with higher scores indicative of greater severity. Severity for the study is the highest score of EXACT-PRO.
Time Frame: Immediately following first IP up to week 56
Population: Full analysis set, baseline EOS>=220/uL
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 202 | 194 | 179
Score on a scale | 51.5 (11.30) | 50.8 (10.70) | 52.0 (11.20)

11. Secondary Outcome: Duration of EXACT-PRO for Patients With Baseline EOS>=220/uL
Description: The EXACT-PRO is a 14-item PRO instrument developed to assess the frequency, severity and duration of COPD exacerbations. Respondents are instructed to complete the electronic diary (eDiary) each evening just prior to bedtime and to answer the questions while onsidering their experiences "today". The daily EXACT-PRO total score has a range of 0-100 with higher scores indicative of greater severity. Event frequency is calculated by comparing the baseline with daily total scores. An increase in EXACT-PRO total score ≥9 for 3 days or ≥12 for 2 days indicate an event has occurred. Calculation of event duration after identification of the following five parameters: 1) onset; 2) three-day rolling average; 3) maximum observed value; 4) threshold for improvement; and 5) recovery. That is, duration of the exacerbation is the time elapse between onset and recovery of the event.
Time Frame: Immediately following first IP up to week 56
Population: Full analysis set, baseline EOS>=220/uL
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 202 | 194 | 179
Days | 82.2 (95.80) | 88.3 (105.30) | 101.7 (113.70)

12. Secondary Outcome: Annual EXACT-PRO Exacerbation Rate Over 56 Weeks Treatment Comparison for Patients With Baseline EOS>=220/uL
Description: The EXACT-PRO is a 14-item PRO instrument developed to assess the frequency, severity and duration of COPD exacerbations. Respondents are instructed to complete the electronic diary (eDiary) each evening just prior to bedtime and to answer the questions while onsidering their experiences "today". The daily EXACT-PRO total score has a range of 0-100 with higher scores indicative of greater severity. Event frequency is calculated by comparing the baseline with daily total scores. An increase in EXACT-PRO total score ≥9 for 3 days or ≥12 for 2 days indicate an event has occurred. Annual EXACT-PRO exacerbation rate is the number of exacerbations per year. Its raw rate is calculated by number of exacerbations divided by the treatment period and then normalized to an annual rate, and is estimated by negative binomial model. Rate ratio between two treatment groups is also estimated through this model.
Time Frame: Immediately following first IP up to week 56
Population: Full analysis set, baseline EOS>=220/uL
Measure: Least Squares Mean (95% Confidence Interval); unit: Exacerbations per year
Arm/Group | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 382 | 378 | 358
Exacerbations per year | 1.14 [0.98 to 1.31] | 1.02 [0.88 to 1.19] | 1.04 [0.90 to 1.21]
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.4080, Negative binomial; Model includes treatment group, EOS cohort, region, background therapy, number of exacerbations in the previous year; Rate ratio = 1.09, 95% CI 2-sided [0.89 to 1.34]
Statistical Analysis 2: Comparison: Benralizumab 100 mg vs Placebo; Test type: Superiority; p = 0.8688, Negative binomial; Model includes treatment group, EOS cohort, region, background therapy, number of exacerbations in the previous year; Rate ratio = 0.98, 95% CI 2-sided [0.80 to 1.21]

13. Secondary Outcome: Number of Participants Having at Least 1 COPD Exacerbation for Patients With Baseline EOS>=220/uL
Description: A COPD exacerbation is defined by symptomatic worsening COPD requiring systemic corticosteroids, antibiotics, or an inpatient hospitalization/death due to COPD.
Time Frame: Immediately following first IP up to week 56
Population: Full analysis set, baseline EOS>=220/uL
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 382 | 379 | 359
Participants | 204 | 203 | 198
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Proportion of participants with >=1 COPD exacerbation; Test type: Superiority; p = 0.4850, Cochran-Mantel-Haenszel; CMH test controlling for EOS cohort, region, and background therapy; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.66 to 1.22]
Statistical Analysis 2: Comparison: Benralizumab 100 mg vs Placebo; Proportion of participants with >=1 COPD exacerbation; Test type: Superiority; p = 0.4489, Cochran-Mantel-Haenszel; CMH test controlling for EOS cohort, region, and background therapy; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.65 to 1.21]

14. Secondary Outcome: Time to First COPD Exacerbation
Description: Time to first COPD exacerbation is from the randomization date to the first occurrence of COPD exacerbation
Time Frame: Immediately following first IP up to week 56
Population: Full analysis set, baseline EOS>=220/uL
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 382 | 379 | 359
Days | 333 [273 to 400] | 329 [262 to 396] | 337 [261 to 390]

15. Secondary Outcome: Annual COPD Exacerbation Rate Associated With ER or Hospitalization Over 56 Weeks Treatment Comparison for Patients With Baseline EOS>=220/uL
Description: Annual COPD exacerbations rate that result in ER or hospitalization is calculated by number of exacerbations resulting ER or hospitalization divided by the treatment period and then normalized to an annual rate, and is estimated by negative binomial model. Rate ratio between two treatment groups is also estimated through this model.
Time Frame: Immediately following first IP up to week 56
Population: Full analysis set, baseline EOS>=220/uL
Measure: Least Squares Mean (95% Confidence Interval); unit: Exacerbations per year
Arm/Group | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 382 | 379 | 359
Exacerbations per year | 0.27 [0.20 to 0.35] | 0.15 [0.11 to 0.20] | 0.25 [0.19 to 0.33]
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.7733, Negative binomial; Model includes treatment group, EOS cohort, region, background therapy, previous year exacerbations associated with hospitalization (Y/N); Rate ratio = 1.06, 95% CI 2-sided [0.73 to 1.53]
Statistical Analysis 2: Comparison: Benralizumab 100 mg vs Placebo; Test type: Superiority; p = 0.0114, Nagative binomial; [statistical method as in outcome 15, analysis 1]; Rate ratio = 0.58, 95% CI 2-sided [0.39 to 0.89]

16. Secondary Outcome: Number of Participants Had COPD-related Healthcare Encounter for Patient With Baseline EOS>=220/uL
Description: Types of healthcare encounter: Hospitalisations (inc. intensive care and/or general care), Emergency department visits, Unscheduled outpatients visits, Home visits, Telephone calls, and ambulance transports.
Time Frame: Immediately following first IP up to week 56
Population: Full analysis set, baseline EOS>=220/uL
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 382 | 379 | 359
Participants
  Hospitalisations | 60 | 38 | 50
  Emergency Department Visits | 36 | 35 | 43
  Unscheduled Outpatient Visits | 219 | 236 | 202
  Home Visits | 18 | 22 | 18
  Telephone calls | 110 | 111 | 104
  Ambulance transports | 16 | 12 | 20

17. Secondary Outcome: Duration of Study Treatment Administration
Description: Duration of study treatment is calculated from first dose date to last dose date + 1 day.
Time Frame: From first dose date to last dose date, 48 weeks per protocol.
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 554 | 552 | 550
Days | 302.4 (85.73) | 304.0 (82.40) | 302.5 (88.47)

18. Secondary Outcome: Serum Concentration of Benralizumab
Description: PK serum samples were collected pre-dose at each visit.
Time Frame: Pre-first dose and pre-dose at end of treatment (week 56)
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Benralizumab 30 mg | Benralizumab 100 mg
Number analyzed (Participants) | 553 | 550
ng/mL
  Baseline: number analyzed (Participants) | 548 | 544
  Baseline | NA (NA) — <LLOQ (Lower limit of quantification) | NA (NA) — <LLOQ (Lower limit of quantification)
  Week 56: number analyzed (Participants) | 375 | 391
  Week 56 | 219.45 (233.21) | 699.89 (243.20)

19. Secondary Outcome: Immunogenicity of Benralizumab
Description: Antidrug antibody (ADA) responses such as ADA prevalence, ADA incidence, ADA persistently positive counts, etc. were presented
Time Frame: Pre-treatment until end of follow-up, week 60 per protocol.
Population: safety analysis set. For each parameter, the number of subjects at risk is to be analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
Number analyzed (Participants) | 554 | 552 | 550
Participants
  ADA prevalence | 53 | 64 | 39
  ADA incidence: number analyzed (Participants) | 547 | 542 | 535
  ADA incidence | 44 | 47 | 24
  Both base/post-baseline positive: number analyzed (Participants) | 547 | 542 | 535
  Both base/post-baseline positive | 5 | 7 | 17
  Only post baseline positive: number analyzed (Participants) | 551 | 547 | 537
  Only post baseline positive | 43 | 46 | 20
  Only baseline positive: number analyzed (Participants) | 550 | 547 | 548
  Only baseline positive | 5 | 11 | 2
  ADA persistently positive: number analyzed (Participants) | 547 | 542 | 535
  ADA persistently positive | 28 | 34 | 14
  ADA transiently positive: number analyzed (Participants) | 547 | 542 | 535
  ADA transiently positive | 15 | 12 | 6
  nAb prevalence | 43 | 43 | 25
  nAb incidence: number analyzed (Participants) | 547 | 542 | 535
  nAb incidence | 41 | 37 | 18

ADVERSE EVENTS:
Time Frame: From the time the patient signed informed consent through the treatment period up to the follow-up visit (week 60).
Arm/Group | Benralizumab 30 mg | Benralizumab 100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 15/554 | 11/552 | 13/550
Serious Adverse Events (participants affected / at risk) | 151/554 | 177/552 | 176/550
Other Adverse Events (participants affected / at risk) | 293/554 | 318/552 | 282/550
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benralizumab 30 mg (N=554) | Benralizumab 100 mg (N=552) | Placebo (N=550)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (3)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1) | 4 (4)
Acute right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0)
Angina unstable (Cardiac disorders) | 2 (2) | 2 (2) | 2 (2)
Aortic valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 8 (8) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (2) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 2 (2) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cor pulmonale chronic (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 4 (4) | 3 (3) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Exomphalos (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (2) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Salivary gland calculus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Atypical mycobacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Atypical mycobacterial lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 3 (3) | 3 (3)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis pharyngeal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 22 (24) | 18 (19) | 16 (16)
Pneumonia bacterial (Infections and infestations) | 5 (5) | 8 (9) | 10 (10)
Pneumonia haemophilus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia moraxella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia necrotising (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Airway burns (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Asbestosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Dural tear (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fractured coccyx (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skin flap necrosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular bypass dysfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram ST-T change (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Non-small cell lung cancer stage IIIB (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 2 (2)
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Monoparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Radicular syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Stupor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Thrombotic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 97 (145) | 78 (101) | 100 (142)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 5 (6)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 4 (5)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin laxity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benralizumab 30 mg (N=554) | Benralizumab 100 mg (N=552) | Placebo (N=550)
Constipation (Gastrointestinal disorders) | 17 (19) | 19 (19) | 15 (17)
Diarrhoea (Gastrointestinal disorders) | 17 (18) | 15 (18) | 6 (7)
Nausea (Gastrointestinal disorders) | 13 (17) | 18 (22) | 13 (15)
Oedema peripheral (General disorders) | 11 (13) | 26 (28) | 11 (11)
Bronchitis (Infections and infestations) | 59 (74) | 84 (113) | 80 (121)
Lower respiratory tract infection (Infections and infestations) | 50 (76) | 32 (47) | 29 (39)
Oral candidiasis (Infections and infestations) | 17 (21) | 13 (18) | 15 (16)
Respiratory tract infection (Infections and infestations) | 10 (10) | 11 (14) | 18 (26)
Respiratory tract infection viral (Infections and infestations) | 15 (21) | 12 (18) | 19 (23)
Sinusitis (Infections and infestations) | 13 (16) | 17 (22) | 20 (22)
Upper respiratory tract infection (Infections and infestations) | 69 (87) | 74 (104) | 65 (97)
Urinary tract infection (Infections and infestations) | 23 (27) | 22 (30) | 15 (22)
Viral upper respiratory tract infection (Infections and infestations) | 83 (126) | 95 (134) | 66 (98)
Back pain (Musculoskeletal and connective tissue disorders) | 21 (23) | 25 (30) | 19 (19)
Headache (Nervous system disorders) | 21 (29) | 26 (30) | 20 (21)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (18) | 14 (20) | 21 (30)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 (30) | 17 (19) | 23 (37)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 (15) | 18 (21) | 13 (17)
Hypertension (Vascular disorders) | 19 (19) | 19 (19) | 18 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
≥ 60 days prior to submission of material for publication/presentation, Institution and PI shall jointly provide AZ with material for review. No publication/presentation may include any of AZ's Confidential Information without AZ's written approval. AZ can request Inst. and PI to withhold material from submission for publication/presentation for an additional 90 days to allow AZ to establish and preserve its proprietary rights in the material being submitted for publication or presentation.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/16/NCT02138916/SAP_000.pdf
  • Study Protocol (2015-07-06): https://cdn.clinicaltrials.gov/large-docs/16/NCT02138916/Prot_001.pdf